CLINICAL TRIAL: NCT01367561
Title: A Phase I Urodynamic Study of the Opioid Antagonist, Naloxone and Intravenous Methylnaltrexone Reverse Opioid Effects on Bladder Function in Healthy Volunteers
Brief Title: Naloxone and Intravenous Methylnaltrexone Effects on Bladder Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, M.D., Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNTX 206
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Healthy Males
MeSH Terms: interventions — Naloxone; methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Naloxone
- Arm 2 (Experimental)
  Interventions: Drug: IV Methylnaltrexone (MNTX)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naloxone
  Arms: Arm 1
Drug: IV Methylnaltrexone (MNTX)
  Arms: Arm 2
Drug: Placebo
  Arms: Arm 3

SUMMARY:
This is a double-blind, randomized, study at a single clinical site investigating the effect of methylnaltrexone and naloxone versus placebo in healthy males who have received a short-acting opioid, remifentanil.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, 18 to 65 yrs with normal urinary function
2. Body weight less than 150 kg and Body Mass Index between 20-32.

Exclusion Criteria:

1. Females
2. History of drug or alcohol abuse
3. History of significant chronic illness (cardiovascular, gastrointestinal, pulmonary, neurologic, endocrine, renal, hepatic, etc.)
4. Subjects who received opioids for one week or longer in the last 2 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-10; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Maximal force of detrusor contraction (Pdet) after administration of MNTX | 14 days
  To investigate the potential benefit of methylnaltrexone in preventing or treating opioid-induced urinary retention.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States